CLINICAL TRIAL: NCT01625520
Title: Mono Centre, Open Label Proof of Concept Study SOM230 in Progressive Medullary Thyroid Cancer Patients and the Combination With RAD001 Upon Progression
Brief Title: SOM230 Alone or in Combination With RAD001 in Patients With Medullary Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Annamaria Colao, Professor, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-023128-26
Record Dates: First submitted 2012-05-25; First posted 2012-06-21 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Medullary Thyroid Cancer
Keywords: Progressive metastatic; postoperative persistent
MeSH Terms: conditions — Carcinoma, Medullary | interventions — pasireotide; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOM230 alone or in combination with RAD001 (Experimental): Patients with progressive metastatic or postoperative persistent medullary thyroid cancer will start the study treatment as a mono therapy with SOM230. Patients benefiting from the treatment will continue with the monotherapy (stable disease or better according to RECIST). Patients progressing will be switched to the combination therapy with SOM230 and RAD001.
  Interventions: Drug: SOM230 alone or in combination with RAD001.

INTERVENTIONS:
Drug: SOM230 alone or in combination with RAD001. — SOM230 (pasireotide) 60 mg i.m. injection once every 28 days, +/- 2 days. RAD001 (everolimus) 10 mg per os daily.

SUMMARY:
A mono centre study to evaluate the efficacy of SOM230 in patients with progressive metastatic or postoperative persistent medullary thyroid cancer.

DETAILED DESCRIPTION:
Medullary thyroid cancer (MTC) is a neuroendocrine tumor originating from thyroid C cells. Neuroendocrine tumors have been demonstrated to express somatostatin receptors as well as mTOR pathway. The somatostatin analogues now available (octreotide and lanreotide) act preferentially through the somatostatin receptor subtype 2 (sst2). In MTC, these compounds have been reported to exert anti-secretive effects on calcitonin but no anti-proliferative effects.SOM230 (pasireotide) is a new somatostatin analogue showing a peculiar binding profile with high affinity for sst1, sst2, sst3, sst5. Preliminary data show SOM230 to be effective in a phase II study on patients with metastatic carcinoid. RAD001 (everolimus) is a novel agent that interacts with mTOR. It was demonstrated to inhibit tumor growth in neuroendocrine tumor cell lines. Some clinical trials have explored the efficacy of a combined therapy with RAD001 plus octreotide in patients with digestive neuroendocrine tumors, highlighting encouraging results in term of tumor control.In particular, octreotide and RAD001 seem to show a synergistic activity in inhibiting neuroendocrine tumor proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with progressive metastatic or postoperative persistent medullary thyroid cancer who have histopathologically confirmed disease and measurable tumor lesions. (Postoperative persistent after surgical removal is characterized by increased levels of calcitonin with or without radiological detectable tumour relapse or metastases.)
* Patients with evidence of biochemical progression of disease, as expressed by progressive increase of serum calcitonin levels, assessed once a month for at least three months before study entry, according to RECIST definitions (elevation of the markers for at least 25 %).
* Disease that is not amenable to surgery, radiation, or combined modality therapy with curative intent.
* Adequate organ function - Karnofsky-Index performance status >60%
* Life expectancy > 6 months
* Age > 18 years
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of randomization and a urine pregnancy test 48 hours prior to the administration of the first study treatment.
* Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary.
* Signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial prior to enrolment.

Exclusion Criteria:

* Unstable systemic diseases including uncontrolled hypertension, active uncontrolled infections, psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Known hypersensitivity to somatostatin analogues.
* Pregnant or breast-feeding patients
* Sign of recurrence of prior or concomitant malignancies (within the last 3 years or requiring active treatment) other than MTC; with the exception of previous basal cell skin cancer, previous cervical carcinoma in situ
* Prior therapy with mTOR inhibitors (e.g. sirolimus, temsirolimus, everolimus)
* Participation in a clinical trial to test an investigational drug within 4 weeks prior to visit 1.
* Any of severe and/or uncontrolled medical conditions:
* Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment,
* QT related exclusion criteria
* Previous treatments with chemotherapy, loco regional therapy (eg, chemoembolization) or interferon are permitted providing that toxicity has resolved to < Grade 1 at study entry and that last treatment was at least 4 weeks prior to baseline assessment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of SOM230 in patients with progressive metastatic or postoperative persistent medullary thyroid cancer | From date of start therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  Efficacy is defined as progression-free survival (PFS), according to RECIST criteria, in patients treated with SOM230.

SECONDARY OUTCOMES:
Efficacy of SOM230 in combination with RAD001 in patients with progressive metastatic or postoperative persistent medullary thyroid cancer. | From date of start therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  Efficacy is defined as progression-free survival (PFS), according to RECIST criteria, in patients treated with SOM230 in combination with RAD001.
Biochemical response | From date of start therapy, 1 month, 2 month, 3 month, 6 month time point evaluation, up to 6 months.
  Biochemical response is defined as the change of calcitonin and carcinoembryonic antigen (CEA) serum concentrations recorded from date of study entry until disease progression compared to baseline. Time-to-biochemical-response is defined as the time from start of the study treatment to first documentation of biochemical response of calcitonin and CEA concentrations, respectively. Duration of biochemical response is defined as the time from the first documentation of biochemical response to the first documentation of biochemical progression or to death due to any cause, whichever occurs first.
Objective tumor response | From date of start therapy, 3 month, 6 month time point evaluation, up to 6 months.
  Objective tumor response (OR) are the overall responses recorded from date of study entry until end of study/study exclusion, according to RECIST definitions, confirmed by repeat measurements. OR includes complete remission (CR), partial (PR), stable disease (SD) and progressive disease (PD) of all measurable tumor lesions of all evaluable patients.
Overall survival | From date of start therapy to the end of the study or death from any cause, whichever came first, up to 6 months.
Time to response | From date of start therapy, 3 month, 6 month time point evaluation, up to 6 months.
  Time to response is defined as the time from start of treatment to the first objective tumor response (PR or CR) observed. Patients who did not achieve a confirmed PR or CR will be censored at last adequate tumor assessment date when they did not progress (including deaths not due to underlying disease)
Duration of response | From time of response to time of tumor progression or death from any cause, whichever came first.
  Duration of response is defined as the time from onset of response (CR/PR) to objective tumor progression or death from any cause. Patients not experiencing progression or death will be censored with the date of their last adequate tumor assessment.
Safety | From date of start therapy until the end of the study, every 30 days, up to 6 months.
  Safety will be evaluated using assessment of adverse events and laboratory data. The assessment of safety will be based on the frequency of adverse events and on the number of laboratory values that are new or worsening based on the common toxicity criteria (CTC) grade. Other safety data (e.g. vital signs) will be considered appropriately.

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, Principal Investigator — "Federico II" University of Naples, Italy
Locations (1):
- Department of Molecular and Clinical Endocrinology and Oncology, "Federico II" University of Naples, Naples, Italy, Italy

REFERENCES:
- [Derived] Faggiano A, Modica R, Severino R, Camera L, Fonti R, Del Prete M, Chiofalo MG, Aria M, Ferolla P, Vitale G, Pezzullo L, Colao A. The antiproliferative effect of pasireotide LAR alone and in combination with everolimus in patients with medullary thyroid cancer: a single-center, open-label, phase II, proof-of-concept study. Endocrine. 2018 Oct;62(1):46-56. doi: 10.1007/s12020-018-1583-7. Epub 2018 Mar 23. PMID 29572709